CLINICAL TRIAL: NCT00403572
Title: A Study of Cerebral-circulatory Response to Intravenous Antihypertensive Treatment in Women With Serious Preeclampsia
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Eldrid Langesæter, MD PhD, Oslo University Hospital
Other Study IDs: ElangeTCD-2006; S-06348b
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Trans cranial Doppler; Cardiac output; systemic vascular resistance; blood pressure
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is a systematical registration of hemodynamic measurements (cardiac output, blood pressure and systemic vascular resistance) in women with serious preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Women with serious preeclampsia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with moderate-to-severe pre-eclapmsia
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Hemodynamic and cerebral-circulatory variations in preeclamptic women | days

CONTACTS AND LOCATIONS:
Overall Officials: Eldrid Langesæter, PhD, MD, Principal Investigator — Oslo University Hospital